CLINICAL TRIAL: NCT00507052
Title: Effect of N-Acetylcysteine on Residual Renal Function in Chronic Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 346147RRF
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Hemodialysis; Renal Failure
Keywords: Hemodialysis; Residual Renal Function
MeSH Terms: conditions — Renal Insufficiency | interventions — Acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine

SUMMARY:
In our opinion, it is worth to check an ability of antioxidant therapy to produce a favorable effect on Residual Renal Function.

The aim of our study is to investigate the effect of N-acetylsysteine on RRF in prevalent HD patients.

DETAILED DESCRIPTION:
Background Preserving residual renal function (RRF) has always been the primary clinical goal for every nephrologists managing patients with chronic kidney disease but not yet on dialysis. RRF in patients on dialysis has proven to be a consistent and powerful predictor of mortality. This is particularly evident for patients treated with peritoneal dialysis (PD): CANUSA study showed that only RRF but not dialysis dose has significant predictive power of mortality [1].

Interestingly, there have been very few studies that have examined the contribution of RRF to outcome in hemodialysis (HD) patients. This is particularly unfortunate because HD patients counts more than 90% of all dialysis population both in Israel and USA. A single study showed that persistence of RRF significantly improved patients' outcome [2].

Moreover, it is well known that RRF deteriorates more rapidly in HD patients than in PD patients [3]. Preservation of RRF remains an unresolved problem in dialysis patients.

The exact mechanism of rapid loss of RRF on HD is not fully understood. Several experimental and clinical studies showed that variety of vascular events and increased oxidative stress in dialysis patients may be due to inhibition of nitric oxide (NO) synthesis by ADMA (Asymmetric Dimethylarginine ), known to be endogenous inhibitor of NO synthetase [4]. ADMA may be significantly reduced by dialysis [5]. Metabolism of ADMA is primarily by the enzyme DDAH , which activity is decreased by inflammation, oxidative stress, diabetes mellitus and hypercholesterolemia [6].

Based on current knowledge, treatment aimed at reducing oxidative stress should decrease ADMA levels [6], and it is logical to suggest that such a therapy might help to preserve RRF in HD patients. In our opinion, it is worth to check an ability of antioxidant therapy to produce a favorable effect on RRF. One preliminary study on effect of antioxidant Vitamin E showed a small beneficial effect on ADMA in chronic kidney disease [7].

N-Acetylcysteine (NAC) is an active antioxidant proved to be safe and beneficial in hemodialysis patents [8]. In our recent study, NAC effectively reduced the ototoxic effect of gentamicin in chronic hemodialysis patients [9].

The aim of our study is to investigate the effect of N-acetylsysteine on RRF in prevalent HD patients.

Methods. Study population. The study will include 20 patients with ESRD, treated with chronic hemo- dialysis in Assaf Harofeh Medical Center.

Patients will be excluded from the study if they are:

1. Patients with acute renal failure
2. Currently treated with antioxidants ( NAC, vitamin E ets.) Study protocol. We planned this study as a prospective cross-sectional study where every patient will serve as his/her own control. Al the patients will continue their previous dialysis and drugs regimen.

After performance of baseline clinical and laboratory examination the patients will receive orally NAC 1200 mg x 2/day for 2 weeks. At the end of this therapy, a follow up PET and Kt/V examination will be performed. These baseline and follow up clinical and laboratory examination will be performed at outpatient basis in our dialysis unit.

The clinical monitoring of all the patients will include:

1. Blood Pressure and Heart Rate - at each of two visits. 2. Review of current medications and doses. 3. Body weight - at each of two visits. 4. Dialysis adequacy: Kt/V 6. Residual renal function examination: 24 hours urinary collection for urea and creatinine and calculation of CCT and residual Kt/V both at baseline and follow up visits.

7. Biochemical studies: ADMA, DDAH, NO - both at baseline and follow up visits.

Statistical analysis The statistical analysis will be performed using the statistical software SPSS-version 10. Parametric data will be expressed as means ± standard deviation and compared by the standard t-test. Non-parametric data will be compared using chi square test. p value of 0.05 or less will be considered significant.

References

1. Bargman J, Thorpe K, Churchill D. Relative contribution of residual renal function and peritoneal clearance to adequacy of dialysis: a reanalysis of the CANUSA study. J Am Soc Nephrol 2001; 12: 2158-62
2. Shemin D, Bostom A, Laliberty P, Dworkin L. Residual renal function and mortality risk in hemodialysis patients. Am J Kidney Dis. 2001; 38: 85-90
3. Moist L, Port F, Orzol S et al. Predictors of loss of residual renal function among new dialysis patients. J Am Soc Nephrol 2000; 11: 556-564.
4. Vallance P, Leone A, Calver A, Collier J, Moncada S. Accumulation of an endogenous inhibitor of nitric oxide synthesis in chronic renal failure.

   Lancet. 1992 Mar 7;339(8793):572-5.
5. Kielstein J, Boger R, Bode-Boger S et al. Asymmetric Dimethylarginine Plasma Concentrations Differ in Patients with End-Stage Renal Disease. J Am Soc Nephrol 1999; 10:594-600
6. Kielstein J, Zoccali C. Asymmetric dimethylarginine: a cardiovascular risk factor and a uremic toxin coming of age? Am J Kidney Dis. 2005;46(2):186-202.
7. Saran R, Novak J, Desai A et al. Impact of vitamin E on plasma asymmetric dimethylarginine (ADMA) in chronic kidney disease (CKD): a pilot study.

   Nephrol Dial Transplant. 2003 Nov;18(11):2415-20.
8. Tepel M, van der Giet M, Statz M et al. The antioxidant acetylcysteine reduces cardiovascular events in patients with end-stage renal failure: a randomized, controlled trial. Circulation. 2003 Feb 25;107(7):992-5.
9. Feldman L, Efrati S, Abramsohn R, Yarovoy I, Gersch E, Eviatar E, Averbukh Z, Weissgarten J. N-Acetylcysteine for prevention of gentamicin-induced ototoxicity in hemodialysis patients. J Am Soc Nephrol 2006; 17 (Suppl): 22A

ELIGIBILITY:
Inclusion Criteria:

* Patients with ESRD, treated with chronic hemodialysis

Exclusion Criteria:

* Patients will be excluded from the study if they are:

  1. Patients with acute renal failure
  2. Currently treated with antioxidants ( NAC, vitamin E ets.)

Ages: 20 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Leonid S Feldman, MD, Principal Investigator — Assaf Harofeh MC
Locations (1):
- Assaf Harofeh, Ẕerifin, Israel